CLINICAL TRIAL: NCT03967197
Title: Is Lidocaine Useful Before Esophageal Manometry and Ambulatory pH Monitoring? A Randomized Controlled Study
Brief Title: Lidocaine Before Esophageal Manometry and Ambulatory pH Monitoring
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-8355
Record Dates: First submitted 2019-05-09; First posted 2019-05-30 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Pain, Acute
Keywords: manometry; pH monitoring; lidocaine
MeSH Terms: conditions — Acute Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Patients randomized to the lidocaine intervention will receive 2 sprays of lidocaine hydrochloride 10% in each nostril 3-5 minutes before their test.
  Interventions: Drug: Lidocaine Hydrochloride
- Placebo (Saline) (Placebo Comparator): Patients randomized to placebo will receive 2 sprays of physiological saline in each nostril 3-5 minutes before their test.
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Saline spray — Physiologic saline spray
  Arms: Placebo (Saline)
Drug: Lidocaine Hydrochloride — Lidocaine hydrochloride 10% spray
  Arms: Lidocaine

SUMMARY:
A randomized controlled trial comparing esophageal manometry and ambulatory pH monitoring test tolerance in the presence versus in the absence of topical lidocaine.

DETAILED DESCRIPTION:
Conventionally, topical nasopharyngeal anesthesia is applied to improve the tolerance of esophageal manometry and ambulatory pH monitoring. However, there is currently no data to support this practice. This randomized controlled trial of lidocaine versus placebo applied before these tests will evaluate the benefit of topical lidocaine anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing esophageal manometry or ambulatory pH monitoring at our center who are able to read and consent to participate in the study.

Exclusion Criteria:

* Patients < 18 years
* Incapacity to provide consent
* History of lidocaine allergy
* Current pregnancy
* Previous esophageal manometry or ambulatory pH monitoring in the last 14 days
* Previous participation in the study
* Severe cirrhosis (Child-Pugh C)
* Severe chronic kidney disease (eGFR<30 mL/min/1.73m2)
* Severe heart failure (New York Heart Association Functional Classification 3-4)
* Severe respiratory failure (dyspnea or oxygen-dependent at rest)
* Any active severe incapacitating chronic or acute medical disease
* Active hospitalization
* Ulcerated, atrophic, infected or recently burned (in the last 30 days) nasopharynx
* Recent surgery involving the nasopharynx (in the last 30 days)
* Severe chronic pain (ex. regular daily use of opioids)
* Previous stroke or any neurological lesion with resulting current sensory deficit
* Major neurocognitive disorder
* Any active severe incapacitating chronic or acute psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Presence of pain during catheter insertion | Assessed once immediately after exam on patient questionnaire
  As reported by patients on a standardized questionnaire

SECONDARY OUTCOMES:
Global patient satisfaction | Assessed once immediately after exam on patient questionnaire
  As reported by patients on a standardized questionnaire (on scale of 1 to 5, 5 being highest satisfaction score)
Presence of other complications during catheter insertion | Assessed once immediately after exam on patient questionnaire
  As reported by patients on a standardized questionnaire
Presence of complications during test recording | Assessed once immediately after exam on patient questionnaire
  As reported by patients on a standardized questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No